CLINICAL TRIAL: NCT02859948
Title: Phase I Open-Label, Sequential Dose Escalation Study Investigating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SKLB1028 When Administered Daily to Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: A Study of SKLB1028 in Subjects With Relapsed/Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1028201601/PRO
Record Dates: First submitted 2016-06-28; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — SKLB1028

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SKLB1028 (Experimental): SKLB1028 capsules in six doses beginning at 20 mg and rising to 200 mg.
  Interventions: Drug: SKLB1028

INTERVENTIONS:
Drug: SKLB1028 — SKLB1028 capsules in six doses beginning at 20 mg and rising to 200 mg.

SUMMARY:
Patients will receive oral SKLB1028 for 28 days to study the side effects, tolerability and best dose for treating relapsed or refractory acute myeloid leukemia With FLT3 Mutations.

DETAILED DESCRIPTION:
It is open-label, dose escalation study designed to characterize the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of orally administered SKLB1028 as a single agent given daily for 28 days. Cohorts of 3 patients receive SKLB1028 until dose limiting toxicity is noted (DLT). At that point cohorts will expand to 6 patients until MTD is determined. Patients not experiencing DLT or significant disease progression could continue receiving SKLB1028 up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be provided.
* Males and females age ≥ 18 years;
* Histopathologically documented primary or secondary AML, as defined by WHO criteria, confirmed by pathology review at treating institution, meeting at least one of the following:

  1. Refractory to at least 1 cycle of induction chemotherapy, or
  2. Relapsed after at least 1 cycle of induction chemotherapy, or
  3. Patient is not, according to the clinical judgment of the Principal Investigator, a candidate for induction chemotherapy due to age, comorbidity, or other factors;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3;
* In the absence of rapidly progressing disease, the interval from prior treatment to time of SKLB1028 administration should be at least 2 weeks for cytotoxic agents, or at least 5 half-lives for noncytotoxic agents;
* Serum creatinine ≤1.5 × ULN;
* Total serum bilirubin ≤ 1.5 × ULN unless considered due to Gilbert's syndrome or leukemic organ involvement;
* Serum AST or ALT ≤ 3.0 × ULN unless considered due to leukemic organ involvement;
* Females of childbearing potential and sexually mature males must agree to use a medically accepted method of contraception throughout the study;

Exclusion Criteria:

* Histologic diagnosis of acute promyelocytic leukemia;
* Clinically active central nervous system leukemia;
* Persistent clinically significant toxicity from prior chemotherapy that is Grade 2 or higher;
* Bone marrow transplant within 100 days prior to study;
* Active, uncontrolled infection;
* Major surgery within 4 weeks prior to study;
* Radiation therapy within 4 weeks prior to study;
* Left ventricular ejection fraction ≤1 × ULN,or﹤50%. Clinically significant ECG QTc prolongation (Male: >450ms, Female: >470ms).Significant cardiac disease.
* Human immunodeficiency virus positivity;
* Active hepatitis B or C or other active liver disease;
* Women who are pregnant, lactating;
* Medical condition, serious intercurrent illness, or other extenuating circumstance that, in the judgment of the Principal Investigator, could jeopardize patient safety or interfere with the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of dose limiting toxicity (DLT)and Adverse Event (AE) | 28 Days

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) | 28 Days
Area under the plasma concentration-time curve (AUC) from time zero to the time point of t (AUC0-tn) | 28 Days
Area under the plasma concentration-time curve (AUC) from time zero to infinity (AUC0-inf) | 28 Days
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 28 Days
Apparent volume of distribution at equilibrium after oral administration（Vss/F） | 28 Days
Plasma Decay Half-Life (t1/2z) | 28 Days
Apparent Oral Clearance (CLz/F) | 28 Days
Average plasma or serum concentration(Cav) | 28 Days
changes in FLT3 mutation status in plasma | 28 Days
Rate of Complete Remission (CR) | 28 Days
Rate of partial remission (PR) | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Ting Liu, Dr., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital，Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No